CLINICAL TRIAL: NCT03037008
Title: Comparison of Perineal Ultrasound in Men Before and After Radical Prostatectomy and in Incontinent Men After Radical Prostatectomy Before and After Operative Treatment With Male Sling
Brief Title: Perineal Ultrasound in Men Before and After Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Winterthur KSW (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-00054
Record Dates: First submitted 2016-08-02; First posted 2017-01-31 (Estimated); Last update posted 2020-04-27 (Actual); Status verified 2019-08

CONDITIONS: Urinary Incontinence, Stress
Keywords: perineal sonography; male sling; post prostatectomy incontinence; ultrasonography
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- continent men after RALP (Active Comparator): perineal sonography, questionnaires, 24h pad tests
  Interventions: Device: Perineal Sonography
- incontinent men after RALP (Active Comparator): perineal sonography, questionnaires, 24h pad tests
  Interventions: Device: Perineal Sonography

INTERVENTIONS:
Device: Perineal Sonography — In a modified lithotomy position (supine position with elevated legs), probands will get an examination of their pelvic floor by using a common ultrasound probe head on the perineum. During the examination, the bladder should be filled with around 300ml. If patient appear with empty bladder, the examination can be repeated on an other date. During the examination, the pelvic floor will be observed during rest, coughing and valsalva-maneuver. One examination takes around 30minutes. During ultrasound, we want to illustrate the urethral mobility, the bladder neck opening and the urethral angle as well as the distance from the urethra to the symphysis.
  Other Names: Perineal Ultrasound

SUMMARY:
Prospective study to evaluate a new technique. Comparison of perineal sonography in men before and after radical prostatectomy and in incontinent men after radical prostatectomy before and after operative treatment with male sling and comparison with pre- and postoperative functional MRI

Inclusion / Exclusion criteria: Inclusion: male, elder than 18years, planned RALP or history of RALP and PPSUI (Post Prostatectomy Stress Urinary Incontinence).

Exclusion: Patients with history of urinary incontinence before radical prostatectomy. Patients with history of radiotherapy in the pelvis. Other diseases involving pelvic floor.

DETAILED DESCRIPTION:
After radical prostatectomy, a part of all patients suffer from urinary incontinence. Until now, only few information exists about the functional anatomy of the male pelvic floor, especially in incontinent men. Transperineal ultrasound is non-hazardous, cheap and easy available method to visualize the pelvic floor and is well established in gynecological examination. literature described the technique of transperineal ultrasound but there are no well established reference lines measured and the number of examined men in the series are small. The investigators want to confirm the published data and probably find new reference lines/parameters, e.g. the distance between the posterior wall of the symphysis to the posterior wall of the urethra in a direct, horizontal line. At the moment, the authors published data about urethral mobility, bladder neck opening and urethral angle. The investigators estimate that there is also a possible significant difference in the distance from the urethra to the symphysis in incontinent men compare to continent men after radical prostatectomy.

Incontinent men can be treated by pelvic floor exercises or, in case of persisting incontinence, with operative treatment. There exists several techniques of implanted slings and meshes, similar to the better known TVT (tension free vaginal tape) in female urinary incontinence, besides the gold standard - the implantation of an artificial sphincter prosthesis. The sling-operations are less invasive, cheaper and preferred by patients du to the fact, that normal micturition is still possible. Nevertheless, around 20% of patients stay incontinent after sling operation. At the moment, it is unknown why they do not profit from the sling. In a previous study functional pelvic cine-MRI in patients with post-prostatectomy incontinence before and after implantation of a bulbourethral composite Suspension were compared. The investigators could find significant differences in the membranous urethral length and could show an elevation oft he bladder neck postoperatively but no significant MRI differences were found between patients showing clinical success or failure. With perineal sonography, the investigators want to establish a prediction tool for sling-operations in patients with urinary stress incontinence after radical prostatectomy.

The purpose of this study is to evaluate whether perineal ultrasound in men is an adequate possibility to evaluate the pelvic floor and its function in the regard of urinary incontinence. The study is trying to find a prediction tool for bulbourethral composite suspension (sling-operation) using transperineal sonography. The investigators further want to establish and confirm parameters/standards to measure the male pelvic floor with the new technique of perineal sonography in men. Further the investigators want to to compare findings from perineal sonography with data from functional MRI in men with urinary incontinence following radical prostatectomy before and after bulbourethral composite suspension. Findings from perineal sonography with results from questionnaires concerning quality of life will be compared.

There is a comparison study with two arms to compare the anatomy and function of the pelvic floor with perineal ultrasound from men prior to RALP due to prostate cancer, without prior history of diseases involving the pelvic floor.

Participants will be asked to participate the study during routine consultations in the department of Kantonsspital Winterthur or selected in our database of the clinical information system searching for radical prostatectomies in the past and recruit these participants by telephone.

In a modified lithotomy position (supine position with elevated legs), probands will get an examination of their pelvic floor by using a common ultrasound probe head on the perineum. During the examination, the bladder should be filled with around 300ml. If patient appear with empty bladder, the examination can be repeated on an other date. During the examination, the pelvic floor is observed during rest, coughing and valsalva-maneuver. One examination takes around 30minutes. During ultrasound, the investigators want to illustrate the urethral mobility, the bladder neck opening and the urethral angle as well as the distance from the urethra to the symphysis.

Urinary incontinence is measured by 24h pad test: Probands have to collect their pads, and scale them before and after using it during 24 hours, to measure the difference. The difference (after-before) shows the amount of lost urine. The results don't have to be exact and a result with a precision of approximately 50ml (= 50g) is acceptable.

Results from urinary analysis (culture) are taken out of medical history from the hospitals database during the period of incontinence to exclude urinary tract infection. If no data is available, urinary analysis will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Male,
* Elder than 18years
* Planned RALP or history of RALP and PPSUI

Exclusion Criteria:

* Patients with history of urinary incontinence before radical prostatectomy.
* Patients with history of radiotherapy in the pelvis.
* Other diseases involving pelvic floor.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
perineal sonography | 1 - 4 weeks before RALP
  In a modified lithotomy position (supine position with elevated legs), probands get an examination of their pelvic floor by using a common ultrasound probe head on the Perineum. During the examination, the pelvic floor is observed during rest, coughing and valsalva-maneuver. Different Parameters (marked Points/anatomical structures) are measured.
IPSS (International Prostate Symptom Score) | 1 - 4 weeks before RALP
  score Points (numeric)
24h pad test | 1 - 4 weeks before RALP
  incontinence is measured by 24 pad test. pads are measured through scales.
perineal sonography | 6 weeks after RALP
  In a modified lithotomy position (supine position with elevated legs), probands get an examination of their pelvic floor by using a common ultrasound probe head on the Perineum. During the examination, the pelvic floor is observed during rest, coughing and valsalva-maneuver. Different Parameters (marked Points/anatomical structures) are measured.
IPSS (International Prostate Symptom Score) | 6 weeks after RALP
  score Points (numeric)
24h pad test | 6 weeks after RALP
  incontinence is measured by 24 pad test. pads are measured through scales.
perineal sonography | 6 months after RALP
  In a modified lithotomy position (supine position with elevated legs), probands get an examination of their pelvic floor by using a common ultrasound probe head on the Perineum. During the examination, the pelvic floor is observed during rest, coughing and valsalva-maneuver. Different Parameters (marked Points/anatomical structures) are measured.
IPSS (International Prostate Symptom Score) | 6 months after RALP
  score Points (numeric)
24h pad test | 6 months after RALP
  incontinence is measured by 24 pad test. pads are measured through scales.
ICIQ SF (International Questionnaire on Urinary Incontinence - Short Form) | 1 - 4 weeks before RALP
  score Points (numeric)
ICIQ SF (International Questionnaire on Urinary Incontinence - Short Form) | 6 weeks after RALP
  score Points (numeric)
ICIQ SF (International Questionnaire on Urinary Incontinence - Short Form) | 6 months after RALP
  score Points (numeric)
IIEF 5 (International Index of Erectile Function) | 1 - 4 weeks before RALP
  score Points (numeric)
IIEF 5 (International Index of Erectile Function) | 6 weeks after RALP
  score Points (numeric)
IIEF 5 (International Index of Erectile Function) | 6 months after RALP
  score Points (numeric)
VAS QoL (Visual Analogue Scale - Quality of Life) | 1 - 4 weeks before RALP
  score Points (numeric)
VAS QoL (Visual Analogue Scale - Quality of Life) | 6 weeks after RALP
  score Points (numeric)
VAS QoL (Visual Analogue Scale - Quality of Life) | 6 months after RALP
  score Points (numeric)
PGI (Patient Generated Index) | 1 - 4 weeks before RALP
  score Points (numeric)
PGI (Patient Generated Index) | 6 weeks after RALP
  score Points (numeric)
PGI (Patient Generated Index) | 6 months after RALP
  score Points (numeric)

CONTACTS AND LOCATIONS:
Overall Officials: Hubert John, Prof., Study Chair — Head of Kantonsspital Winterthur Urology
Locations (1):
- Kantonsspital Winterthur, Winterthur, Switzerland

IPD SHARING:
Plan to Share IPD: No